CLINICAL TRIAL: NCT03248908
Title: Pupillary Dilation Reflex Assessment for Intraoperative Analgesic Titration [PUP-AIT]. A Double Blinded Randomized Trial.
Brief Title: Pupillary Dilation Reflex Assessment for Intraoperative Analgesic Titration.
Acronym: PUP-AIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Principle investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17/28/319
Record Dates: First submitted 2017-08-01; First posted 2017-08-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Anesthesia
Keywords: pupillary reflex; nociception; heart rate; intraoperative monitoring
MeSH Terms: conditions — Acute Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, the performer of the pupillary reflex measurement, and the postoperative health care provider are masked for the study arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1 (Experimental): Pupillary dilation reflex based perioperative intravenous remifentanil administration. Starting dose 5 ng/ml by continous infusion, dosage adjustments are made after pupillary dilation reflex assessment every 10 minutes. When PPI score is 1, the dosage is decreased with 0.2 ng/ml. When PPI score is greater than 1, the dosage is increased with 0.2 ng/ml.
  Interventions: Diagnostic Test: Pupillary dilation reflex
- Intervention 2 (Active Comparator): Anesthesiologist based perioperative intravenous remifentanil administration (daily practice, standard of care). Starting dose 5 ng/ml, dosage adjustments are made when deemed necessary by attending anesthesiologist.
  Interventions: Other: Standard of care
- Intervention 3 (Experimental): Pupillary dilation reflex based perioperative intravenous sufentanil administration. Starting dose 0.1 mcg/kg bolus, dosage adjustments are made after pupillary dilation reflex assessment every 10 minutes. When PPI score is 1, no supplementary administration is executed. When PPI score is greater than 1, a supplementary bolus of 0.1 mcg/kg is given.
  Interventions: Diagnostic Test: Pupillary dilation reflex
- Intervention 4 (Active Comparator): Anesthesiologist based perioperative intravenous sufentanil administration (daily practice, standard of care). Starting dose 0.1 mcg/kg bolus, dosage adjustments are made when deemed necessary by attending anesthesiologist.
  Interventions: Other: Standard of care

INTERVENTIONS:
Diagnostic Test: Pupillary dilation reflex — Perioperative pupillary dilation reflex assessment is executed every 10 minutes from start sedation until extubation in patients allocated to study arm Intervention 1 and Intervention 3
  Arms: Intervention 1; Intervention 3
Other: Standard of care — Perioperative opioid administration based on the attending anesthesiologist decision (mainly including assessment of heart rate, blood pressure, and limb movement)
  Arms: Intervention 2; Intervention 4

SUMMARY:
In this double blinded randomized controlled study, the pupillary dilation reflex is used for as a nociceptive indicator for opioid administration during elective surgery under general anesthesia.

DETAILED DESCRIPTION:
An infrared camera of the video pupillometer measures the pupillary dilation reflex (PDR) in response of a nociceptive stimulus. This autonomic reflex, parasympathetic mediated in sedated patients, can be generated by various pain stimuli (built in standardized protocol, surgical incision, …) The PDR is a robust reflex, even in patients under general anesthesia, and provides a potential evaluation of the autonomous circuit within the nociceptive evaluation based on pupil dilation upon A-delta and C fibers in both electrical or mechanic stimulation. This double blind randomized controlled trial involving American Society of Anesthesiologists (ASA) classification I-III patients undergoing elective surgery under general anesthesia are recruited. Enrolled patients are randomized in four groups: (1) remifentanil administration depending on PDR results, (2) remifentanil administration depending on decision attending anesthesiologist, (3) sufentanil administration depending on PDR results, (4) sufentanil administration depending on decision attending anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* > 18 jaar
* Elective abdominal or gynaecological operation
* ASA (American Society of Anesthesiologists classification): I - II - III

Exclusion Criteria:

* History of invasive ophthalmological surgery
* Known bilateral eye disease
* Known optical of oculomotor nerve deficit
* Active psychiatrical disease
* Proven active pheochromocytoma
* Opioid usage > 7 days preoperative
* Ongoing oncological treatment with chemotherapeutic agents
* Usage of A-1 adrenergic of beta-blocking agents
* Preoperative usage of benzodiazepines
* Topical atropine or phenylephrine (eye droplets)
* Planned perioperative usage of dopamine antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | From patient extubation until postoperative day 5
  Numeric rating scale (NRS) pain assessment
Postoperative analgesia | From patient extubation until postoperative day 5
  Analgetic consumption

SECONDARY OUTCOMES:
Stimulation intensity to elicit PDR | From the day of surgery at the start of general anesthesia, assessed every 10 minutes until the end of surgery or extubation, whichever came first, assessed up to 4 hours
  Necessary stimulation intensity generated by the pupillometer to elicit a PDR
Baseline pupil diameter | From the day of surgery at the start of general anesthesia, assessed every 10 minutes until the end of surgery or extubation, whichever came first, assessed up to 4 hours
  Pupil size before stimulation
Pupillary dilation reflex amplitude | From the day of surgery at the start of general anesthesia, assessed every 10 minutes until the end of surgery or extubation, whichever came first, assessed up to 4 hours
  The amplitude of the pupil enlargement after nociceptive stimulation
Pupillary pain index (PPI) | From the day of surgery at the start of general anesthesia, assessed every 10 minutes until the end of surgery or extubation, whichever came first, assessed up to 4 hours
  Generated PPI score by the pupillometer in accordance to given stimulation and pupillary dilation reflex amplitude
Opioid usage during surgery | From the day of surgery at the start of general anesthesia, assessed every 10 minutes until the end of surgery or extubation, whichever came first, assessed up to 4 hours
  Total dose remifentanil or sufentanil administrated during surgery, in microgram
Extubation time | From the day of surgery at the termination of propofol infusion until patient extubation, assessed up to 2 hours
  The time between stop of propofol administration and patient extubation, in minutes
Postoperative nausea and vomiting | From patient extubation until postoperative day 5
  Frequency of nausea or vomiting after surgery, in numbers of events
Length of stay at the postanesthesia care unit | From admission at the postanesthesia care unit until discharge to the nursing ward, assessed up to 24 hours
  Hours of admission at the postanesthesia care unit after surgery until discharge to the nursing ward, in minutes
Length of hospital stay | From the day of the planned surgery until hospital discharge, assessed up to 5 days
  Length of hospital stay, in days
Postoperative health status | From extubation until 1 month after surgery
  Assessed by 5-level EQ-5D version (EQ-5D-5L), quality of life and health status questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Davina Wildemeersch, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vlaenderen DV, Hans G, Saldien V, Wildemeersch D. Pupillary reflex dilation and pain index evaluation during general anesthesia using sufentanil: a double-blind randomized controlled trial. Pain Manag. 2022 Nov;12(8):931-941. doi: 10.2217/pmt-2022-0027. Epub 2022 Oct 3. PMID 36189668